CLINICAL TRIAL: NCT06058091
Title: A Multicenter Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of RY_SW01 Cell Injection Therapy in Systemic Sclerosis
Brief Title: RY_SW01 Cell Injection Therapy in Systemic Sclerosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Renocell Biotech Company (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Sun Lingyun, MD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RYSW202301
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Systemic Sclerosis
Keywords: RY_SW01 cell injection
MeSH Terms: conditions — Scleroderma, Systemic | interventions — macrophage-derived immunosuppressor factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase II-Placebo group (Placebo Comparator): Receive the best basic treatment
  Interventions: Drug: Basic treatment
- Phase II-low-does group (Experimental): Receive the best basic treatment and a million cells per kilogram of body weight
  Interventions: Drug: RY_SW01 cell injection; Drug: Basic treatment
- Phase II-high does group (Experimental): Receive the best basic treatment and two million cells per kilogram of body weight
  Interventions: Drug: RY_SW01 cell injection; Drug: Basic treatment

INTERVENTIONS:
Drug: RY_SW01 cell injection — Administer basic treatment with an injection of RY_SW01 cell solution
  Other Names: UC-MSC treatment
  Arms: Phase II-high does group; Phase II-low-does group
Drug: Basic treatment — Basic treatment for SSc
  Other Names: immunosuppressor

SUMMARY:
Systemic sclerosis (SSc) tends to progress to involve multiple vital organs within 5 years of diagnosis, significantly impacting patient prognosis and survival. Clinical indications suggest that early intervention is more favorable for long-term outcomes in patients. Although guidelines recommend various drugs for symptomatic treatment, there is currently no standard therapy or effective medication to slow the progression of the disease. Therefore, for patients with diffuse SSc, as defined by a skin score of 10≤mRSS≤30 points, who have been treated with at least two therapies, including steroids, immunosuppressive agents, biologics, etc., within 5 years of diagnosis, the applicant intends to develop a drug that can both modulate the immune system and counteract fibrosis. The goal is to provide long-term benefits to patients through early intervention.

DETAILED DESCRIPTION:
This clinical trial is a multicenter Phase I/II clinical trial, which includes two stages: Phase I dose-escalation and Phase II dose-expansion. The Phase I dose-escalation stage adopts a single-arm trial design, aiming to explore the safety, tolerability, and preliminary efficacy of RY_SW01 cell injection in treating patients with systemic sclerosis. The Phase II dose-expansion stage adopts a randomized, double-blind controlled trial design, intending to explore the safety, efficacy, and changes in disease-related biomarkers of RY_SW01 cell injection in treating systemic sclerosis patients.

Based on the characteristics of this product and pre-clinical study data, as well as integrating the safety and efficacy data of similar types of drugs and clinical trials for the same or similar indications published domestically and internationally, the researchers and sponsors jointly selected the trial exploration doses as low dose 1.0×10^6 cells/kg and high dose 2.0×10^6 cells/kg.

The trial will enroll systemic sclerosis patients aged ≥18 and ≤65 years, who must meet all inclusion criteria and none of the exclusion criteria. Approximately 81-87 subjects are planned to be enrolled to undergo dose-escalation and dose-expansion trials with RY_SW01 cell injection. The dose-escalation stage plans to enroll 6-12 evaluable subjects, and the dose-expansion stage plans to enroll 75 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form.
2. Aged between 18 and 65 years (inclusive), regardless of gender.
3. Diagnosed with systemic sclerosis (SSc) based on the 2013 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria for SSc.
4. Screened as diffuse cutaneous SSc patients with a disease duration of ≤5 years (disease onset defined as the time of the initial diagnosis of SSc).
5. Previously treated with at least two of the following therapies: corticosteroids, immunosuppressants, biologic agents, and others, and have a skin score of 10≤mRSS≤30 points.

Exclusion Criteria:

1. At screening, subjects with a forced vital capacity (FVC) predicted percentage <50%.
2. Previously diagnosed with pulmonary arterial hypertension or, at rest, had a mean pulmonary arterial pressure >25mmHg measured by right heart catheterization or had a systolic pulmonary artery pressure >45mmHg measured by echocardiography at screening.
3. Presence of clinical symptoms requiring hospitalization for one of the following conditions at screening, whether newly occurring or worsening of pre-existing symptoms within 6 months: myocardial infarction, stroke, renal crisis, severe uncontrolled hypertension (≥160/100mmHg); or within 3 months: unstable ischemic heart disease, uncontrolled arrhythmia, heart failure (New York Heart Association III/IV stage), left ventricular ejection fraction <50% as indicated by echocardiography, renal insufficiency, or hypertensive crisis as judged by the investigator.
4. Concurrent autoimmune connective tissue diseases other than systemic sclerosis, with the exception of patients with secondary Sjögren's syndrome.
5. Presence of any of the following laboratory abnormalities at screening:

   1. Hematology abnormalities: Hemoglobin <100g/L; White blood cell count <3.0×109/L; Neutrophil absolute count <1.5×109/L; Platelet count <100×109/L.
   2. Hepatic function abnormalities: ALT or AST >3 times the upper limit of normal (ULN); Total bilirubin >3 times ULN.
   3. Renal function abnormalities: Estimated glomerular filtration rate (eGFR) <60mL/min/1.73m2 or any clinically significant laboratory abnormalities that may affect the interpretation of study data or the subject's participation in the study as determined by the investigator.
6. Positive testing for human immunodeficiency virus (HIV) antibody, active syphilis, active hepatitis C (positive HCV antibodies and positive HCV-RNA), HBsAg positive and HBV-DNA positive at screening; history of severe active bacterial, viral, fungal, parasitic, or other infections during the screening period.
7. Receipt of live vaccines/attenuated vaccines within 2 months prior to enrollment.
8. Occurrence of any of the following within 3 months prior to enrollment: a. Major trauma or major surgery (including joint surgery) or anticipated major surgery during the study, which the investigator believes would pose an unacceptable risk to the subject. b. Plasma exchange or extracorporeal photopheresis treatment. c. Participation in any other clinical trials.
9. Prior treatment with stem cell-related drugs.
10. History of any malignancy within the past 5 years prior to enrollment, except for adequately treated or excised basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical carcinoma.
11. Intolerance or contraindication to the study treatment, including any of the following: a. Allergy to albumin contained in the investigational product excipient. b. Lack of suitable peripheral venous access.
12. History of smoking, alcohol abuse, or drug abuse within the past 12 months or during the screening period:

    1. Smoking defined as an average daily consumption of ≥5 cigarettes within the 3 months prior to screening.
    2. Alcohol abuse defined as consuming more than 14 units of alcohol per week (1 unit of alcohol = 350ml of beer, or 45ml of spirits, or 150ml of wine) within the 3 months prior to screening.
    3. Drug abuse defined as having a history of drug abuse.
13. Plans for conception during the trial period until at least 1 year after cell infusion, unwillingness to use effective contraceptive measures with their partners, or plans for sperm or egg donation.
14. Deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 24 weeks
Change of mRSS | 24 weeks

SECONDARY OUTCOMES:
Change in mRSS from baseline | 12 weeks
Change in lung function (FVC predicted percentage) from baselineRY_SW01 cell injection. | 24 weeks
Proportion of subjects with treatment failure. | 24 weeks
Proportion of subjects showing improvement in mRSScell injection (Improvement defined as a decrease in mRSS from baseline by ≥25%). | 24 weeks
Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) from baseline to 24 weeks after RY_SW01 cell injection. | 24 weeks
Biological markerTGF-β, VEGF, TNF-a, and Th17 cell subset proportions from baseline to 12 and 24 weeks after RY_SW01 cell injection. | 12weeks 24weeks
  TNFR1, anti-Scl-70 antibodies, IL-6, TGF-β，TNF-a,Th17

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, Study Director — Jiangsu Renocell Biotech Company
Locations (1):
- Department of Rheumatology and Immunology, Nanjing Drum Tower Hospital, the Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No